CLINICAL TRIAL: NCT03292770
Title: EFFICACY STUDY OF THE UTILIZATION OF A FLUSHING CATHETER FOR REMOVAL OF CERVICAL MUCUS BEFORE AN EMBRYO TRANSFER: A RANDOMIZED PILOT CONTROLLED TRIAL
Brief Title: Mucus Removal Before Embryo Transfer
Acronym: MUCRET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Jorge Rodriguez-Purata, Dr. Jorge Rodriguez-Purata, Fundacion Dexeus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMD-CAT-2017-01
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Infertility; Embryo Transfer
Keywords: Embryo Transfer; Flushing catheter; Pregnancy rate; Frozen Embryo Tranfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: All participants will be randomized by an intention to treat approach. All other components of the IVF/ICSI cycle including stimulation medications, monitoring protocols, etc. will be at the discretion of the participant's primary physician; while this information will be documented it will not constitute criteria for enrolment. The group allocation will take place the day of the embryo transfer. The clinician will randomize all included patients into one of the two study groups using an open computer-generated list.
Who Masked: Participant, Outcomes Assessor
Masking Description: All included patients will be blinded of the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Embryo transfer will be performed as per clinic's routine protocol, where cervical mucus is gently removed with a cotton swab. No manipulation of the cervical canal is executed.
- Flushing Group (Experimental): A catheter will be used to perform a flushing of the cervical canal with culture media. The Flushing Catheter has a flared proximal end that is designed to affix to a standard Luer slip syringe and a pre-curved distal closed end, with a biseled opening on the side, 2mm from the tip, in which liquid flushes towards the outside of the cervical canal.
  Device: Cook Flushing Catheter J-IUIC-352200 (3.5fr 20cm flushing catheter with positioner closed end) (CEE approval).
  Interventions: Device: Flushing Catheter

INTERVENTIONS:
Device: Flushing Catheter — A catheter will be used to performed a flushing of the cervical canal with culture media.
  Arms: Flushing Group

SUMMARY:
Despite these revolutionary changes in the laboratory, little has changed with the process of embryo transfer (ET). A study to prospectively evaluate the role of cervical mucus removal prior to embryo transfer on pregnancy rates in ART will be undertaken.

DETAILED DESCRIPTION:
ET involves placing the embryo(s) obtained before assisted reproduction technology (ART) into the uterus via a catheter advanced through the cervical canal. Yet this is the final, and in some respects the most critical, process in the sequential events that encompass an ART cycle. If an embryo cannot be delivered to the uterine cavity atraumatically and in a location for optimal implantation, the steps of ovarian hyperstimulation, oocyte retrieval, embryo culture, and embryo selection will have no benefit. Contamination of the catheter with blood may be a marker for difficult ET and has also been linked to poor ET outcomes. When retrospectively assessing outcomes, Goudas et al. (1) demonstrated a clinical pregnancy rate of 50% with no blood, and this rate fell by half when a small amount of blood was noted on the catheter tip. Pregnancy rates fell even further, to 10%, when there was a significant amount of blood (1). Similarly, in a preliminary study, blood or mucus on the tip was associated with a significantly lower pregnancy outcome (2). Blood and mucus were associated with an increased risk for unsuccessful transfers with odds ratios of 1.9 and 1.8, respectively. Although all these data suggest a possible role of cervical mucus in embryo transfer, there is no clinical evidence on the effect of removal of cervical mucus on the outcome of IVF/ICSI. In view of this uncertainty, a study to prospectively evaluate the role of cervical mucus removal prior to embryo transfer on pregnancy rates in ART will be undertaken. It is hypothesized that removal of cervical mucus will achieve higher clinical pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* IVF or OD patients with supernumerary embryos (oocyte's age will be considered as patient's age).
* Normal transvaginal ultrasound at screening, without evidence of clinically significant abnormality consistent with finding adequate for ART with respect to uterus and adnexa
* Single embryo transfer
* Embryo transfer at the blastocyst stage
* Embryo with a morphological classification of ≥3BB

Exclusion Criteria:

* Preimplantation genetic diagnosis and/or screening

Max Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 1118 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate | 20 days after embryo transfer
  Defined as the proportion of patients with a gestational sac seen 20 days after embryo transfer

SECONDARY OUTCOMES:
Biochemical Pregnancy Rate | 9 days after embryo transfer
  Defined as the proportion of patients with ≥25 mIU/L of serum βhCG 9 days after embryo transfer
Early Pregnancy Loss Rate | 20 days after embryo transfer
  Defined as the proportion of patients with a pregnancy loss following a positive pregnancy test and/or a detectable gestational sac

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Rodriguez-Purata, MD, Principal Investigator — Hospital Universitario Dexeus
Locations (1):
- Hospital Universitario Dexeus, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided